CLINICAL TRIAL: NCT05211102
Title: Venous Sinus Thrombosis : Clinical Picture and Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam medhat edward, Mariam medhat edward, Assiut University
Other Study IDs: Venous sinus thrombosis
Record Dates: First submitted 2022-01-25; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Vein Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral venous sinus thrombosis (cvst) is an underdiagnosed neurological condition with variable clinical presentations and variable risk factors CVST is often an underdiagnosed cause of acute or slowly progressive neurological deficit.

With increasing awareness of the entity and easy accessibility to the non-invasive test like CT and MRI scans,CVST cases are now being diagnosed more frequently and it is now thought to occur more commonly than previously assumed.it is also probably true that this condition is more frequent in underdeveloped countries

ELIGIBILITY:
Inclusion Criteria:

1. All patients admitted to the neurology department and ER of an assuit university hospital with the diagnosis of venous sinus thrombosis
2. accepting to participate in the study
3. of both sex above 18 years and below 70 years

Exclusion Criteria:

* 1. any case evident to have neurological deficit due to cause other than venous sinus thrombosis 2. patients refused to participate in this study 3-patients with uncertainty about her imaging study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sex above 18years and below 70years presenting to Assiut University Hospital with cerebral venous sinus thrombosis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
cerebral venous sinus thrombosis | 1 year
  Clinical presentations of cerebral venous sinus thrombosis

IPD SHARING:
Plan to Share IPD: Undecided